CLINICAL TRIAL: NCT02360709
Title: A Prospective, Multi-center, Single-arm Observational Registry Trial Evaluating the Safety and Efficacy of CRE8 Sirolimus-Eluting Stent in the Treatment of Patients With De Novo Coronary Artery Lesions
Brief Title: Safety and Efficacy of the CRE8 Sirolimus-Eluting Stent for the Treatment of De Novo Coronary Artery Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CID S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRE8-China-SA
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CRE8 group: CRE8 sirolimus-eluting stent
  Interventions: Device: CRE8 sirolimus-eluting stent

INTERVENTIONS:
Device: CRE8 sirolimus-eluting stent — The CRE8 stent system consists of a sirolimus eluting coronary stent firmly held on the distal end of a semicompliant balloon catheter. This stent is made of cobalt chromium alloy and is coated with a thin carbon film.The outer surface of the stent has dedicated grooves for containing the pharmaceutical formulation, which is composed of the drug sirolimus and a mixture of long chain fatty acids.

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and deliverability of the CRE8 sirolimus-eluting stent system in the treatment of patients with de novo coronary artery lesions.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm observational registry trial planned to enroll 800 subjects. All 800 subjects enrolled will receive CRE8 stents. Clinical follow-up will be performed at 1 month, 6 months,12 months and annually up to 5 years after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 75 years, male or female without pregnancy;
* Patients with clinical evidence of asymptomatic heart disease, stable or unstable angina, or old myocardial infarction;
* De novo lesions of native coronary arteries;
* Target vessel diameter between 2.25mm and 4.5 mm, and target lesion length ≤ 60mm by visual estimation;
* Target lesion diameter stenosis ≥ 70% by visual estimation;
* Each target lesion must be implanted the same stent (CRE8);
* Patients is eligible for percutaneous coronary intervention (PCI) and is an acceptable candidate for surgical revascularization (CABG);
* Patients with left ventricular ejection fraction ≥40%;
* Patients who can understand the nature of the study, agree to participate and accept angiographic and clinical follow-up, and have provided written informed consents.

Exclusion Criteria:

* Patients with acute myocardial infarction (AMI) within 72 hours;
* Chronic total occlusion lesion (TIMI flow 0 before procedure), Left main disease and/or triple-vessel lesion that might require treatment;
* Heavily calcified or tortuous lesions which cannot be successfully pre-dilated, and lesions which are not suitable for stent delivery and deployment;
* In-stent restenosis;
* Thrombotic lesions;
* Patients who had received any other stent in the past one year;
* Patients with acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl);
* Patients with cardiogenic shock, acute infection, known bleeding or coagulation disorder, or with a history of active gastrointestinal bleeding, ulcer, cerebral hemorrhage or subarachnoid hemorrhage and stroke within 6 months;
* Patients who allergic to aspirin, clopidogrel, ticagrelor, ticlopidine, heparin, contrast agent, sirolimus, polymer, Co-Cr alloy, or with contraindication to aspirin or clopidogrel or ticagrelor;
* Patients with life expectancy less than 1year;
* Patients who had participated in another investigational drug or device trial that has not completed the primary endpoint;
* Patient is in the opinion of the investigator, unable to comply with the requirements of the study protocol;
* Patients who had underwent heart transplant surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This trial plans to enroll 800 subjects with de novo coronary artery lesions. Patients with reference diameter between 2.25mm and 4.5 mm (by visual estimation) and lesion length not more than 60mm (by visual estimation) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF,device-oriented endpoint) | 12months after the procedure

SECONDARY OUTCOMES:
Target lesion failure (TLF,device-oriented endpoint) | 1month,6months,2years,3years,4years and 5years follow-up
The patient-oriented composite endpoint includes all-cause death, all MIs, or any revascularizations | 1month,6months,12months and annually up to 5years follow-up
Stent thrombosis per ARC definition | 1month,6months,12months and annually up to 5years follow-up
device and lesion success rates | immidiately after the procedure
clinical success rate | 7 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, MD, Principal Investigator — Fu Wai Hospital, National Center for Cardiovasular disease
Locations (1):
- Fuwai Hospital,National Center for Cardiovasular disease, Beijing, Beijing Municipality, China